CLINICAL TRIAL: NCT03461913
Title: Can Shorter Time Intervals Help the Baby Survive the Triad Effect of Maternal Hypertension, Caesarean Section and Spinal Anesthesia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 32
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Neonatal Hypoxia and Asphyxia
MeSH Terms: conditions — Asphyxia Neonatorum; Asphyxia | interventions — Cesarean Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal pregnancy (Active Comparator): women at full term healthy pregnancy who underwent elective Cesarean section
  Interventions: Procedure: Cesarean section
- pregnancy hypertension (Active Comparator): women at full term pregnancy associated with hypertension who underwent elective Cesarean section
  Interventions: Procedure: Cesarean section

INTERVENTIONS:
Procedure: Cesarean section — Lower segment elective Cesarean section
  Other Names: Elective Cesarean section

SUMMARY:
Patients were classified into two equal groups using the presence or absence of hypertension during pregnancy into: hypertensive group (BP>140/90) and normotensive group (BP≤140/90. The surgical time intervals are assessed and classified the patients accordingly into short and log time interval subgroups (induction of regional anesthesia to delivery (I-D), initial skin incision to delivery (S-D), and uterine incision to delivery (U-D)

DETAILED DESCRIPTION:
Surgical times components; induction of regional anesthesia till delivery (I-D interval); incision of the skin till delivery (S-D interval); and incision of the uterus till delivery (U-D interval)) were recorded using a stopwatch.

Immediately after delivery, umbilical cords were clamped on both ends and an arterial blood sample was collected anaerobically in a pre-heparinized insulin syringe. PH, base excess (BE), carbon dioxide pressure (PCO2), Oxygen pressure (PO2) and Bicarbonate (HCO3) levels were measured at 37oC by pH and gas analyzer (Gem, Premier3000, USA). The gas analysis was done in less than 30 minutes after sampling.

Apgar score was assessed by a neonatologist at the 1st and 5th minutes after birth . Advanced resuscitation included positive pressure ventilation, chest compression and/or drugs administration. All resuscitated babies were transferred to neonatal intensive care unit for post resuscitation care. Fetal distress was defined by an umbilical cord pH <7.12

ELIGIBILITY:
Inclusion Criteria:

* full term pregnancy
* singleton pregnancy
* no medical disorders except hypertension in group 2

Exclusion Criteria:

* Multiple pregnancies
* complicated pre-eclamptic cases as placental abruption, eclampsia or HELLP syndrome,
* preterm pregnancies,
* true knots of the cord
* reduced liquor,
* in labour patients,
* fetal distress
* infants with major congenital malformations

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-10-29 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
umbilical cord Ph | immediately after delivery
  umbilical cords were clamped on both ends and an arterial blood sample was collected anaerobically in a pre-heparinized insulin syringe

SECONDARY OUTCOMES:
Apgar score | 1 and 5 minutes after delivery
  assessment of Appearance, Pulse, Grimace, Activity, and Respiration

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided